CLINICAL TRIAL: NCT04502498
Title: Preoperative Detection of Subclinical Lower Limb Deep Venous Thrombosis in Locally Advanced Bladder Cancer Patients Candidate for Radical Cystectomy
Brief Title: Preoperative Subclinical DVT Screening in Locally Advanced Bladder Cancer Patients Candidate for Radical Cystectomy.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Samer Morsy, Urology lecturer, Kasr El Aini Hospital
Other Study IDs: Cairo University Hospital
Record Dates: First submitted 2020-08-04; First posted 2020-08-06 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Bladder Cancer Patients Candidate for Radical Cystectomy
MeSH Terms: interventions — Echocardiography, Doppler

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 60 patients with local advanced bladder cancer: Local advanced bladder cancer patients candidate for radical cystectomy
  Interventions: Diagnostic Test: Lower limb duplex & doppler

INTERVENTIONS:
Diagnostic Test: Lower limb duplex & doppler — Lower limb duplex and doppler one week before radical cystectomy

SUMMARY:
Preoperative subclinical DVT screening in locally advanced bladder cancer patients candidate for radical cystectomy.

DETAILED DESCRIPTION:
60 patient with local advanced bladder cancer are subjected to preoperative lower limb duplex within 1 week preoperative to radical cystectomy

ELIGIBILITY:
Inclusion Criteria:

* any age
* Any sex
* Muscle invasive bladder cancer local advanced patients candidate for radical cystectomy

Exclusion Criteria:

* Unfit patients
* any contraindication for surgery
* obese
* coagulopathy
* bedridden

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Locally advanced Bladder cancer patients candidate for radical cystectomy and with no symptoms of DVT
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Preoperative subclinical DVT | 6 months
  Asymptomatic patients candidate for radical cystectomy